CLINICAL TRIAL: NCT06138119
Title: The Impact of Gender Stereotypes on Fiberoptic Intubation Performance: A Randomized Controlled Simulation Study
Brief Title: The Impact of Gender Stereotypes on Fiberoptic Intubation Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: V.K.V. American Hospital, Istanbul (Other)
Responsible Party: Principal Investigator, Murat Tümer, MD, Principal Investigator, V.K.V. American Hospital, Istanbul
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: GenderAndFob
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Stereotype-threat; Intubation; Difficult or Failed; Gender
Keywords: Gender Stereotype; Fiberoptic Intubation
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Intervention Model Description: It will be a 2x2 between-subject factorial design. Simulation FOE (Fiberoptic Intubation) scores will be the dependent variable. Being male or female and stereotype threat will be the study's independent variables. There will be four groups to be compared: Male anesthesiologists in the experimental group (1), male anesthesiologists in the control group (2), female anesthesiologists in the experimental group (3), female anesthesiologists in the control group (4).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Female anesthesiologists in the experimental group (Experimental): Stereotype threat manipulation will be performed on the female anesthesiologist in the experimental group just before they are taken into the testing room.
  Interventions: Behavioral: stereotype threat manipulation
- Female anesthesiologists in the control group (No Intervention): The female anesthesiologists in the control group will not be given any prior information.
- Male anesthesiologist in the experimental group (Experimental): Stereotype threat manipulation will be performed on the male anesthesiologist in the experimental group just before they are taken into the testing room.
  Interventions: Behavioral: stereotype threat manipulation
- Male anesthesiologist in the control group (No Intervention): The male anesthesiologists in the control group will not be given any prior information.

INTERVENTIONS:
Behavioral: stereotype threat manipulation — Stereotype threat is the thought that a person will be negatively evaluated and judged regarding a negative stereotype that belongs to the group to which he/ she belongs. Stereotype threat manipulation will be performed on the male and female participants in the experimental group just before they are taken into the testing room. For manipulation, the following sentences will be said to the participants in the experimental group: "We aim to compare fiberoptic intubation performance between male and female anesthesiologists. Additionally, we are investigating whether the high inclination of males towards computer games has any impact on their fiberoptic intubation success." The other participants (Control Group) will not be given any prior information.
  Arms: Female anesthesiologists in the experimental group; Male anesthesiologist in the experimental group

SUMMARY:
Gender bias and stereotypes have been recognized as pervasive factors influencing various aspects of society, including professional settings. Within the realm of medical practice, understanding the potential impacts of such biases on performance is of paramount importance. Anesthesiology, a field that demands technical precision, teamwork, and rapid decision-making, is not immune to the potential effects of gender stereotypes on performance outcomes. This study aims to explore the potential influence of gender stereotype manipulation and stereotype threat on the fiber-optic intubation (FOE) performance of female anesthesiology residents.

Stereotype threat refers to the apprehension individuals experience when their actions or abilities are evaluated within the context of negative stereotypes associated with their social group. Such threat has been shown to adversely affect cognitive and motor performance in various domains. In medical education, where skills are honed through training, understanding the role of stereotype threat is crucial to fostering equitable learning environments and ensuring patient safety.

ELIGIBILITY:
Inclusion Criteria:

1.Residents in the Department of Anesthesiology and Reanimation at Hacettepe University Faculty of Medicine, who have completed their initial year of residency and have prior experience in FOE.

Exclusion Criteria:

1. Not meeting the above criteria
2. Not willing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Fİberoptic Intubation (FOE) Performance | During FOE simulation
  Change in FOE scores in the experimental group compared to the control group. Measurements were conducted on the ORSIM Bronchoscopy simulator using its own measurement parameters, including Task Completion Time (s), Collision Avoidance (%), and Final Score (min 0-100). A decrease in task completion time, an increase in collision avoidance percentage, and a higher final score indicate that the participant performed fiberoptic intubation more effectively.

CONTACTS AND LOCATIONS:
Locations (1):
- VKV Amerikan Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: at the and of the study

REFERENCES:
- [Background] Steele CM, Aronson J. Stereotype threat and the intellectual test performance of African Americans. J Pers Soc Psychol. 1995 Nov;69(5):797-811. doi: 10.1037//0022-3514.69.5.797. PMID 7473032
- [Background] Hall WJ, Chapman MV, Lee KM, Merino YM, Thomas TW, Payne BK, Eng E, Day SH, Coyne-Beasley T. Implicit Racial/Ethnic Bias Among Health Care Professionals and Its Influence on Health Care Outcomes: A Systematic Review. Am J Public Health. 2015 Dec;105(12):e60-76. doi: 10.2105/AJPH.2015.302903. Epub 2015 Oct 15. PMID 26469668
- [Background] Ankay Yilbas A, Canbay O, Akca B, Uzumcugil F, Melek A, Calis M, Vargel I. The effect of playing video games on fiberoptic intubation skills. Anaesth Crit Care Pain Med. 2019 Aug;38(4):341-345. doi: 10.1016/j.accpm.2018.11.012. Epub 2018 Dec 21. PMID 30579943
- See also: Fiberoptic simulation device — http://www.orsim.com